CLINICAL TRIAL: NCT02065349
Title: A Phase 2a Enriched Enrollment Randomized Withdrawal Study to Assess Analgesic Efficacy and Safety of ASP8477 in Subjects With Peripheral Neuropathic Pain
Brief Title: A Study Into Pain Relief Given by ASP8477 for Peripheral Neuropathic Pain (Either Post-herpetic Neuralgia or Painful Diabetic Peripheral Neuropathy) and Its Safety
Acronym: MOBILE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8477-CL-0020; 2013-002521-27 (EudraCT Number)
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Post-Herpetic Neuralgia (PHN); Neuropathic Pain; Painful Diabetic Peripheral Neuropathy (PDPN)
Keywords: peripheral neuropathy; PHN; pain; PDPN
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia; Peripheral Nervous System Diseases; Pain | interventions — ASP8477

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): oral
  Interventions: Drug: Placebo
- ASP8477 (Active Comparator): oral
  Interventions: Drug: ASP8477

INTERVENTIONS:
Drug: ASP8477 — oral
  Arms: ASP8477
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the painkilling efficacy of ASP8477 relative to mock (placebo) in patients that have been diagnosed with painful diabetic peripheral neuropathy or postherpetic neuralgia determined by the change in the average daily pain intensity in patients that initially respond favorably to treatment with ASP8477.

DETAILED DESCRIPTION:
The study will consist of a Screening Period, Single-Blind Treatment Period, Double-Blind Randomized Withdrawal Period and Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* PDPN subject must have:

  * Established diagnosis of diabetes (type I or II) with painful diabetic peripheral neuropathy and glycosylated hemoglobin (HbA1c) ≤ 11% at Screening.
  * Stable glycemic control (HbA1c ≤ 11%) achieved by a drug regimen for at least 3 months prior to Screening.
  * At least a 1-year history of DPN pain.
  * Diabetic distal symmetrical polyneuropathy symptoms (including pain) stable for at least the last 3 months prior to Screening based on PI judgment and subject-reported medical history.
* PHN subject must have pain present ≥ 6 months after healing of the herpes zoster rash.

Exclusion Criteria:

* Subject has significant pain of an etiology other than PDPN or PHN, or clearly non differentiated pain, or plantar fasciitis, heel spurs, tibial neuropathy, Morton's neuroma, bunions, metatarsalgia, arthritis in feet, ischemic pain, neurological disorders unrelated to diabetic neuropathy, skin condition in area of neuropathy that could alter sensation, malignancy, or current orthostatic hypotension, hypo or hypertension, syncope or clinically significant ECG, clinical intolerance to Non-steroidal anti-inflammatory drugs (NSAIDs) or ASP8477, depression, psychosis or psychiatric or neurological illness, BMI of over 35, renal impairment or failure, alcohol (ETOH) or drug abuse, GI complaints.
* Previous investigational therapy within 28 days or 5 half lives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2015-02-13 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Change in mean of 24-hour average pain intensity, Numeric pain rating scale (NPRS) | Baseline of the double-blind randomized withdrawal period to the last 3 days of double-blind randomized withdrawal period

SECONDARY OUTCOMES:
Time to treatment failure | Date of randomization to first 3 consecutive days of double-blind period with an observed treatment failure
  Treatment failure is defined as mean 24 hour pain intensity was equal or more than 4 with at least a 30% increase in pain intensity relative to baseline of the double-blind randomized withdrawal period
Responder rate to ASP8477 in the Single-Blind Period | Baseline of the single-blind period (last 3 days of the placebo run-in period) to baseline of the double-blind period (last 3 days of the single-blind period
Patient Global Impression of Change (PGIC) score | From the baseline of the single-blind period to End of Treatment Visit (Day 49 or upon early discontinuation)
Safety assessed by TEAE and SAE, laboratory tests, vital signs, C-SSRS, PWC and MWC scores, Bond-Lader score | From Screening to End of Study Visit (13 weeks)
  TEAE=Treatment Emergent Adverse Events, SAE = Serious Adverse Event, C-SSRS = Columbia Suicide Severity Rating Scale, PWC = Physician Withdrawal Checklist, MWC = Marijuana Withdrawal Checklist
Composite of pharmacokinetics of ASP8477 concentration: Trough concentration (Ctrough), observed maximum concentration (Cmax), Area under the curve (AUC)0-6 | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Europe B.V.
Locations (17):
- Czechia (6):
  - Site: CZ42003, Choceň
  - Site: CZ42004, Litomyšl
  - Site: CZ42011, Olomouc
  - Site: CZ42014, Prague
  - Site: CZ42001, Rychnov nad Kněžnou
  - Site: CZ42002, Slezská Ostrava
- Germany (2):
  - Site: DE49003, Cologne
  - Site: DE49005, Neuss
- Poland (5):
  - Site: PL48003, Bialystok
  - Site: PL48004, Poznan
  - Site: PL48001, Poznan
  - Site: PL48002, Torun
  - Site: PL48005, Warsaw
- United Kingdom (4):
  - Site: GB44001, Glasgow, Scotland
  - Site: GB44003, Ipswich
  - Site: GB44006, London
  - Site: GB44002, Manchester

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=217